Title: Influence of the Sleep Pattern in Patients Submitted to Bariatric Surgery

**NCT number:** 03485352

**Date:** 03/04/2021

## **INFORMED CONSENT FORM**

You are being invited to participate in the research entitled "Influence of sleep pattern and chronotype of metabolic, anthropometric and biochemical responses in patients undergoing bariatric surgery", under the responsibility of the researchers: Aline Cunha Carvalho and Cibele Aparecida Crispim. The Informed Consent Form will be obtained by the researcher Aline Cunha Carvalho. In their participation, researchers will analyze their information related to medical and nutritional care after performing bariatric surgery. This analyzed information will be related to what you reported to the clinic nutritionist in your appointments, about your eating habits (what you eat, times and places); what the nutritionist evaluated from his body measurements, such as weight, waist, hip and neck circumferences. Percentages of lean body fat will also be evaluated; blood tests (collection of 3 ml) and polysomnography data (tests performed by medical request). Polysomnography is an indicated test that analyzes the sleep pattern in a very detailed way. The research team will apply questionnaires to answer you about sleeping habits (what time do you sleep, if you are sleepy, how do you evaluate your sleep) and also about your chronotype (time of day you prefer to do your activities). The risks are that during the blood collection, it may be painful for the volunteer, resulting in bruises ("purx") and / or swelling caused by blood collection, embarrassment (" shame") for weight measurement and body circumferences and during the application of questionnaires. Every care will be taken to avoid any such occurrence. For measurements of weight and body circumferences it will be performed in an exclusive room for this purpose. The application of questionnaires will be done in a way that does not constrain or repress any reported information, seeking to establish trust between the volunteer and the research team. In order to perform blood collection in this study, it will be carried out under the responsibility of laboratories with extensive experience in this activity. The benefit will be a description for science of possible associations between sleep habits and chronotype and the response to weight loss in patients undergoing bariatric surgery, which may favor the success of this type of treatment for obesity. There is a risk of being identified, but care will be taken to prevent this from happening. In order to minimize this risk for the participant, all questionnaires to be filled out will be coded with numbers and in none of them will the individual's name be described. The results of the research will be published as soon as possible, and even so, your identity will be preserved. You will have no financial expense and gain from participating in the survey. You are free to stop participating in the survey at any time without any harm or duress. An original copy of this Informed Consent Form will spin with you. Any questions, you can contact:

Cibele Aparecida Crispim. Adjunct Professor I, Nutrition Course, Faculty of Medicine, Federal University of Uberlândia. Address: Avenida Pará, 1720- Bloco 2U, Sala 20, Campus Umuarama. Phone: 3218-2084.

Aline Cunha Carvalho. Postgraduate in Health Sciences, Faculty of Medicine, Federal University of Uberlândia. Address: Avenida Pará, 1720 Block 2U, room 20. Campus Umuarama. Phone: 3218-2389.

You can also contact the Ethics Committee on Research with Human Beings - Federal University of Uberlândia: Av. João Naves de Ávila, n° 2121, block A, room 224, Campus Santa Mônica - Uberlândia - MG, CEP: 38408-100; phone: (34) 3239-4131.